CLINICAL TRIAL: NCT03219996
Title: Risk Factors Influenced Prognosis of Acute Fulminant Myocarditis by Analyzing Clinical Characteristics and Complications, Laboratory Findings, Treatments, and Electrocardiographic and Echocardiographic Data.
Brief Title: Risk Factors for Predictors of In-hospital Death in Acute Fulminant Myocarditis
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: myocarditis20161226
Record Dates: First submitted 2017-07-04; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Viral Myocarditis; Cardio-Renal Syndrome; Risk Factor, Cardiovascular
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-survivor group
  Interventions: Other: prognosis
- survivor group
  Interventions: Other: prognosis

INTERVENTIONS:
Other: prognosis — The participants were divided into two groups based on survival at their hospital discharge.

SUMMARY:
The investigators performed a retrospective, single-center observational study, and the participants with acute fulminant myocarditis were included.Then, the investigator analyzed the risk factors of in-hospital death in these participants with acute fulminant myocarditis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of acute fulminant myocarditis

Exclusion Criteria:

chronic renal dysfunction refuse medical treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The definition of a fulminant acute myocarditis was the presence of a rapid onset of aggressive life-threatening disease accompanied by cardiogenic shock with multiple organ dysfunction syndrome, acute severe heart failure, fatal arrhythmias, high-degree atrioventricular blockade, or sudden cardiac death following a flu-like illness.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Renal Impairment Influence Prognosis of Acute Fulminant Myocarditis | 2017-01-30

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjun Yang, PhD, Principal Investigator — First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: Undecided